CLINICAL TRIAL: NCT05475405
Title: Scapulo-Thoracic Mobilization Compared to IASTM in Patients With Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01073 Iqra
Record Dates: First submitted 2022-07-24; First posted 2022-07-26 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Mechanical Neck Pain
Keywords: IASTM; scapulo-thoracic mobilization; mechanical neck pain

STUDY DESIGN:
Intervention Model Description: 32 Participants were recruited in the study and divided into two groups. Group A was given intervention Scapulothoracic mobilization and Group B with IASTM.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scapulothoracic mobilization along with conventional physical therapy for mechanical neck pain. (Experimental): conventional physical therapy:
  Scapulothoracic mobilization:
  Patient in prone lying position. The left hand of the physical therapist lifts the scapula to distract from the thoracic wall while the right hand mobilizes and stretches the inferior muscle groups attached to the scapula.
  Interventions: Other: scapulothoracic mobilization
- IASTM with conventional physical therapy for mechanical neck pain (Active Comparator): Conventional Physical Therapy:
  IASTM (Instrument Assisted Soft Tissue Technique):
  Patient sitting or prone lying Restrictions and myofascial adhesions assessed prior to treatment fanning strokes at 45 degree angles to skin be applied using the tool
  Interventions: Other: IASTM

INTERVENTIONS:
Other: scapulothoracic mobilization — Patient in prone lying position. The left hand of the physical therapist lifts the scapula to distract from the thoracic wall while the right hand mobilizes and stretches the inferior muscle groups attached to the scapula.
  Arms: Scapulothoracic mobilization along with conventional physical therapy for mechanical neck pain.
Other: IASTM — Restrictions and myofascial adhesions should be assessed prior to treatment along both sides using IASTM tool and a lubricant.
  Once restrictions are assessed, fanning strokes at 45 degree angles to skin should be applied using the tool. This technique should be performed for 20 seconds parallel to the muscle fibers and 20 seconds perpendicular to the muscle fibers for each muscle group in scapulothoracic region. Total time for IASTM application is 10 mints. Upon completing all this patient should be given a home plan consisting of 2 different self-stretches targeting levator scapulae and upper trapezius
  Other Names: Instrument assisted Soft tissue mobilization.
  Arms: IASTM with conventional physical therapy for mechanical neck pain

SUMMARY:
SCAPULO-THORACIC MOBILIZATION COMPARED TO IASTM IN PATIENTS WITH MECHANICAL NECK PAIN

DETAILED DESCRIPTION:
Mechanical neck pain is common musculoskeletal condition that causes work disabilities and is not self-limiting. One of the main causes for mechanical neck pain is forward head posture, which is common and but not ideal posture adopted by many workers and students who presents with head being anterior to the shoulder. Imbalances in the normal muscle function reported in such patients with inhibited deep neck flexors, serratus anterior and rhomboids and tightened pectoralis, upper trapezius and levator scapula.

Neck and scapula have some common muscle attachments and abnormal loads on cervical or thoracic spine change the biomechanics of muscles present in these regions, which eventually cause trigger points Management of scapulo-thoracic joint focuses on correcting posture, restoring flexibility of the scapula including the pectoralis minor, levator scapulae, rhomboids, mobilization and soft tissue techniques.

IASTM is ergonomically designed stainless steel tool, and has recently gained much popularity for elevating pain, reducing trigger points and improving ROMs because it has deeply penetrating power as compared to mobilization through hand. This technique works by both along the mobilizing muscle fibers or parallel to the muscle fibers.

ELIGIBILITY:
Inclusion Criteria:

* Age group 18 to 40 years
* Both gender groups
* Non radiating neck pain

Exclusion Criteria:

* History of cervical and thoracic spine surgery
* Vertibro-basilar insufficiency
* Sign of serious pathology like malignancy
* Signs of systemic inflammatory disorder
* Patient with diagnosed hypertension
* (scapular area pathology)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 3 weeks
  Changes from baseline Numeric pain Rating Scale is used to objectively assess musculoskeletal pain as marked by the patient. It is a 10 point scale from 0 to 10. 0 depicts no pain at all and 10 shows worst pain ever felt. It was measured at baseline, at 3rd session after 6th weeks of the intervention.
NDI (neck disability index) | 3 weeks
  The questionnaire has 10 items concerning pain and activities of daily living including personal care, lifting, reading, headaches, concentration, work status, driving, sleeping and recreation. The measure is designed to be given to the patient to complete, and can provide useful information for management and prognosis of those with neck pain
Goniometer | 3 weeks
  goniometer is a device that measures an angle or permits rotation of an object to a definite position

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No